CLINICAL TRIAL: NCT02276092
Title: Effectiveness of a Regional Antimicrobial Stewardship Program to Reduce the Length of Stay of Patients Admitted to Hospital With Community-acquired Pneumonia: a Pragmatic Multi-centre Clinical Study
Brief Title: Impact of a Regional Antimicrobial Stewardship on the Length of Stay of Patients Admitted to Hospital With Pneumonia
Acronym: RASPCAP
Status: Completed | Type: Observational
Sponsor: Royal Victoria Hospital, Canada (Other)
Responsible Party: Principal Investigator, Giulio DiDiodato, principal investigator, Royal Victoria Hospital, Canada
Other Study IDs: RASP2013
Record Dates: First submitted 2014-10-22; First posted 2014-10-27 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pneumonia
Keywords: Community-acquired pneumonia; Pragmatic study; Multi-center; Time-dependent bias; antimicrobial stewardship; prospective audit and feedback
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Antimicrobial Stewardship

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- intervention: exposure to antimicrobial stewardship intervention
  Interventions: Other: antimicrobial stewardship
- control: usual care with no exposure to antimicrobial stewardship

INTERVENTIONS:
Other: antimicrobial stewardship — A member of the antimicrobial stewardship program will prospectively review the patient's medical record and make recommendations to the most responsible physician in the care of that patient
  Other Names: prospective audit and feedback
  Groups: intervention

SUMMARY:
This study evaluates the effectiveness of an antimicrobial stewardship program to reduce the length of stay of patients admitted to hospital with a diagnosis of pneumonia. The antimicrobial stewardship program will be implemented in several hospitals in Ontario, Canada. The program will identify patients with pneumonia, review their charts and make recommendations to their attending physicians about antibiotic management.

DETAILED DESCRIPTION:
Antimicrobial stewardship is defined as any activity that promotes the appropriate selection, dosing, route and duration of antibiotic therapy. Antimicrobial stewardship programs usually include pharmacists and/or doctors with expertise in infection diseases management. Prospective chart review and physician feedback is a common intervention used by antimicrobial stewardship programs to improve antibiotic utilization and patient outcomes.

Pneumonia is the most common reason for antibiotic utilization in hospitals. Significant variation in antibiotic utilization for patients with pneumonia has been repeatedly demonstrated in published studies despite the existence of best-practice treatment guidelines. Treatment variation from these guidelines has been demonstrated to result in worse outcomes such as increased mortality. Antimicrobial stewardship programs can help reduce the treatment variation from guidelines.

Despite improvements in certain outcomes, antimicrobial stewardship programs have not demonstrated any impact on the length of stay of patients admitted to hospital with pneumonia. Part of this absence of evidence may be due to poor study design and failure to recruit sufficient patients. This study will include the implementation of an antimicrobial stewardship program across many hospitals and the study design and analysis will account for the design problems of the previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Community-acquired pneumonia
* Immunocompetent
* Age > 18 years

Exclusion Criteria:

* Admitted to an intensive care unit or high intensity unit
* Requiring invasive or non-invasive ventilation
* Life expectancy less than 3 months
* Hospitalization within the previous 3 months for at least 48 consecutive hours
* Immunocompromised defined as defined as having leukemia, lymphoma, HIV with CD4 count <=200, splenectomy or on cytotoxic chemotherapy
* Neutropenic [defined as a PMN count<=0.5x109 cells/L] from any cause
* Receiving immunosuppressants [defined as >=40 mg prednisone daily (or steroid equivalent) for >=2 weeks preceding hospitalization OR any other immunosuppressant used for systemic illness OR to prevent transplant rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over the age of 18 years admitted to a hospital ward with a diagnosis of community-acquired pneumonia as determined by the most responsible physician
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Days from time of admission to time of discharge from hospital to a maximum of 14 days from the date of admission (or time to censoring at 14 days from the date of admissionor competing event depending on which comes first)
  Time (measured in days) from date of admission to one of the following potential outcomes, discharge alive, censoring at 14 days post admission, death, admission to an intensive care unit, or transfer to another hospital

SECONDARY OUTCOMES:
Days of antibiotic therapy | Days of antibiotic therapy for the treatment of pneumonia measured from the first day of antibiotic administered to the final day of antibiotic administered upto a maximum of 80 days
  Total days of antibiotics administered for the treatment of community-acquired pneumonia
Mortality rate | 30 day post-discharge from hospital
  Deaths that occur post-discharge from hospital up to 30 days post-discharge
Readmission to hospital | 30 day post-discharge from hospital
  Readmissions to hospital that occur post-discharge from hospital up to 30 days post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Giulio DiDiodato, MD, Principal Investigator — Physician
Locations (1):
- Royal Victoria Regional Health Centre, Barrie, Ontario, Canada